CLINICAL TRIAL: NCT04059393
Title: Impact of a PCRC-Supported Legacy Intervention in Pediatric Palliative Care
Brief Title: PCRC-Supported Legacy Intervention in Pediatric Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Palliative Care Research Cooperative Group (Network)
Responsible Party: Principal Investigator, Terrah Akard, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC PED 14130; NCI-2019-05051 (Registry Identifier: NCI, Clinical Trials Reporting Program); R01NR015353 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Care Giver; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (web-based legacy intervention) (Experimental): Patients participate in a web-based legacy intervention by answering questions about themselves and uploading videos, photographs, and music to create a digital story within 2 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (standard of care) (Active Comparator): Patients receive standard of care. Patients have the option to participate in the web-based legacy intervention after 2 months.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Complete web-based legacy intervention
  Arms: Group I (web-based legacy intervention)
Other: Best Practice — Receive standard of care
  Arms: Group II (standard of care)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a web-based legacy intervention works in improving the quality of life in caregivers and younger patients with cancer that has come back (recurrent) or does not respond to treatment (refractory). Legacy-making, defined as doing or saying something to be remembered, may reduce the suffering of children with cancer and their caregivers. Currently, there is little information about what kinds of legacy-making activities are helpful from the perspective of children. Using a web-based digital storytelling intervention, this study may help researchers examine what children think about these legacy-making activities and what kinds of activities might be helpful to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the impact of legacy-making on coping strategies and adjustment outcomes among children with refractory or relapsed cancer.

II. To examine the impact of legacy-making on coping strategies and adjustment outcomes among parent caregivers.

III. To examine the process of implementing a web-based legacy-making intervention for children with refractory or relapsed cancer and their parent caregivers by obtaining parent self-reports (e.g., What did you and your child-like/not like about the intervention? How difficult was it to complete the intervention? What made it difficult? What else you would like to teach us?).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in a web-based legacy intervention by answering questions about themselves and uploading videos, photographs, and music to create a digital story within 2 weeks.

GROUP II: Patients receive standard of care. Patients have the option to participate in the web-based legacy intervention after 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-17 years will be included so the sample will reflect similar developmental understandings that death is permanent and universal. Ages 18 and up are excluded because they begin very different developmental stages of independence as they often leave home and begin college and careers. The principal investigator (PI) or trained clinical trials associate (CTA) will determine the primary parent caregiver by gathering objective information (e.g., number of hours spent per week with the child) from the child's legal guardian during the initial recruitment process
* Relapsed or refractory cancer disease states: This will be determined by parent self-report. This determination will be made at any point within the illness trajectory
* Able to speak, understand, read, and type English: Participants will be limited to those who meet this criterion because the instruments and methods proposed in this research have not been translated in foreign languages
* Participants will be limited to those who have internet access to allow us to successfully examine the feasibility of a web-based intervention
* Absence of cognitive impairment: Cognitive impairment will be determined by the PI or CTA during the consent process. If the child or parent does not understand the consent process (e.g., does not understand project goal, does not understand study procedures), the PI or CTA will gently conclude the recruitment process. Any data already collected will not be included in data analysis, and the participant will be considered withdrawn

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Child coping strategies | Change between baseline and 2 months post-baseline.
  Will be measured using the Response to Stress Questionnaire (RSQ). The 57 items are rated from 1-4 indicating frequency of responses to stress, resulting in 5 factors: (a) primary control coping, (b) secondary control coping, (c) disengagement coping, (d) involuntary engagement, and (e) involuntary disengagement. The total score is the total sum of all 57 items, ranging from 57-228. The 5 factor scores are computed as the sum of the appropriate subscales.
Child adjustment | Change between baseline and 2 months post-baseline.
  Will be measured using 27-item Pediatric Quality of Life (PedsQL) Inventory Cancer Module to assess child quality of life. We used Child Self-Report versions for ages 5-7, 8-12, and 13-17. Parents completed Parent Proxy-Reports. Items for 7-year-olds were rated on a 3-point Likert scale. Items for children aged 8-17 years and parents were rated on a 5-point Likert scale. Multidimensional scales include pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, and communication. Scores are transformed to a 0-100 scale. To calculate scores by dimensions, the mean score = sum of the items over the number of items answered. The total score is the sum of all the items over the number of items answered on all the scales. Higher scores indicate lower problems.
Child adjustment | Change between baseline and 2 months post-baseline.
  Will be measured using the Parent-Adolescent Communication Scale (PACS) to assess parent-child communication. Children and parents complete 20-40 items to assess parent-child communication. A total score is calculated ranging from 20-100 with higher scores indicating more positive communication.
Parent adjustment | Change between baseline and 2 months post-baseline
  Will be measured using the Parent-Adolescent Communication Scale (PACS) to assess parent-child communication. Children and parents complete 20-40 items to assess parent-child communication. A total score is calculated ranging from 20-100 with higher scores indicating more positive communication.
Parent adjustment | Change between baseline and 2 months post-baseline.
  Will be measured using the Adult Self-Report (ASR). The 126-item ASR will assess adaptive functioning and problems. Items are rated on a 3-point Likert scale. Scores in relation to norms for each gender and age are based on national probability samples. Higher scores indicate the item is true for the individual.
Parent coping strategies | Change between baseline and 2 months post-baseline
  Will be measured using the Response to Stress Questionnaire (RSQ). The 57 items are rated from 1-4 indicating frequency of responses to stress, resulting in 5 factors: (a) primary control coping, (b) secondary control coping, (c) disengagement coping, (d) involuntary engagement, and (e) involuntary disengagement. The total score is the total sum of all 57 items, ranging from 57-228. The 5 factor scores are computed as the sum of the appropriate subscales.

SECONDARY OUTCOMES:
Parent satisfaction | Up to 3 months
  Will be measured using a Follow-up Parent survey that includes multiple choice and open-ended questions related to intervention benefits and suggestions for future research. Counts and frequencies will be reported for parent responses to multiple choice questions. Responses to open-ended questions will undergo thematic content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Terrah Akard, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitlow ML, Gilmer MJ, Dietrich MS, Cho E, Akard TF. Digital Stories Created by Children With Advanced Cancer. J Pediatr Hematol Oncol Nurs. 2024 Sep-Oct;41(5):336-348. doi: 10.1177/27527530241267296. Epub 2024 Sep 10. PMID 39257031
- [Derived] Foster Akard T, Dietrich MS, Friedman DL, Wray S, Gerhardt CA, Given B, Hendricks-Ferguson VL, Hinds PS, Cho E, Gilmer MJ. Effects of a Web-Based Pediatric Oncology Legacy Intervention on Parental Coping. Oncol Nurs Forum. 2021 May 1;48(3):309-316. doi: 10.1188/21.ONF.309-316. PMID 33855995
- [Derived] Robson PC, Dietrich MS, Akard TF. Associations of Age, Gender, and Family Income with Quality of Life in Children With Advanced Cancer. J Pediatr Oncol Nurs. 2021 Jul-Aug;38(4):254-261. doi: 10.1177/1043454221992321. Epub 2021 Mar 9. PMID 33686901
- [Derived] Akard TF, Dietrich MS, Friedman DL, Wray S, Gerhardt CA, Hendricks-Ferguson V, Hinds PS, Rhoten B, Gilmer MJ. Randomized Clinical Trial of a Legacy Intervention for Quality of Life in Children with Advanced Cancer. J Palliat Med. 2021 May;24(5):680-688. doi: 10.1089/jpm.2020.0139. Epub 2020 Sep 30. PMID 32996842
- [Derived] Akard TF, Wray S, Friedman DL, Dietrich MS, Hendricks-Ferguson V, Given B, Gerhardt CA, Hinds PS, Gilmer MJ. Transforming a Face-to-Face Legacy Intervention to a Web-Based Legacy Intervention for Children With Advanced Cancer. J Hosp Palliat Nurs. 2020 Feb;22(1):49-60. doi: 10.1097/NJH.0000000000000614. PMID 31804281